CLINICAL TRIAL: NCT00845299
Title: An Open-Label, Randomized, Phase 2 Study of the Effects of Artificial Tears Preserved With Benzalkonium Chloride (AT-BAK) on the Response to the Latanoprost Punctal Plug Delivery System (L PPDS) in Subjects With Ocular Hypertension (OH) or Open-Angle Glaucoma (OAG)
Brief Title: Study of the Effects of Artificial Tears on the Response to the Latanoprost Punctal Plug Delivery System in Subjects With Ocular Hypertension or Open-Angle Glaucoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPL GLAU 04
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: glaucoma; ocular hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Benzalkonium Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Latanoprost punctal plug and use of artificial tears containing Benzalkonium Chloride
  Interventions: Drug: Latanoprost punctal plug; Drug: artificial tears preserved with Benzalkonium Chloride
- 2 (Experimental): Latanoprost punctal plug only
  Interventions: Drug: Latanoprost punctal plug

INTERVENTIONS:
Drug: Latanoprost punctal plug — Control of IOP compared to baseline for the experimental dose of Latanoprost punctal plug for 6 weeks or until loss of efficacy.
Drug: artificial tears preserved with Benzalkonium Chloride
  Arms: 1

SUMMARY:
The purpose of this study is to determine the effect of artificial tears preserved with Benzalkonium Chloride (AT-BAK) on the IOP response to the L-PPDS and to evaluate the safety of the L-PPDS in subjects with OH or OAG following treatment.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years with ocular hypertension or open-angle glaucoma
* Subjects who have a best-corrected visual acuity of 20/100 or better

Exclusion Criteria:

* Subjects who wear contact lenses
* Uncontrolled medical conditions
* Subjects with a known sensitivity to latanoprost, BAK, or any other products required for the study
* Subjects requiring chronic topical artificial tears, lubricants, and/or requiring any other chronic topical medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
IOP change from baseline | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Cuzzani, MD, Study Director — QLT Inc.
Locations (1):
- Menlo Park, California, United States